CLINICAL TRIAL: NCT00236626
Title: A 9 Month, Double-Blind, Placebo-Controlled Study With a Blinded Crossover Transition to Open-Label Extension, Evaluating the Safety and Effectiveness of Topiramate on Insulin Sensitivity in Overweight or Obese Type 2 Diabetes Patients
Brief Title: A Study of the Safety and Effectiveness of Topiramate on Insulin Sensitivity in Overweight or Obese Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003715
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-04

CONDITIONS: Obesity; Diabetes Mellitus, Type 2; Diabetes Mellitus, Adult-Onset
Keywords: Type 2 Diabetes; Obesity; Insulin Resistance; Body Mass Index; Hypertension; Hyperlipidemia; Sulfonylurea; Topiramate; Adult-Onset Diabetes Mellitus; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Insulin Resistance; Hypertension; Hyperlipidemias; Metabolic Syndrome | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to investigate (1) the effect of topiramate on insulin sensitivity in overweight or obese patients with type 2 diabetes mellitus and (2) the safety of topiramate in type 2 diabetic patients. The study will also investigate the effect of topiramate on body weight, body fat, fat distribution, and metabolic control including both glucose and lipid levels.

DETAILED DESCRIPTION:
Topiramate is not approved for the treatment of obesity. This double-blind, placebo controlled study investigates the effect of topiramate on insulin sensitivity in overweight or obese patients with Type 2 Diabetes. After a screening phase, patients are randomized to receive either topiramate (96 milligrams[mg] twice daily) or placebo for 9 months in the double-blind phase. After 9 months, patients have the option to continue in the open-label phase and receive treatment with topiramate for 1 year. Patients in the placebo group then receive topiramate with dosage increasing gradually to 96 mg twice daily, with the option of increasing to 256 mg twice daily. Patients in the topiramate group continue with the maintenance dose received during the double-blind phase, with the option of increasing to 256 mg twice daily. Assessments of effectiveness made monthly include insulin sensitivity, body composition (as measured by computed tomography [CT]), body weight and Body Mass Index (BMI), waist and hip circumferences, fasting lipid profile, fasting glucose and hemoglobin type A1c (HbA1c) levels, and blood pressure. Safety evaluations, including incidence of adverse events, clinical laboratory results, vital signs, and electrocardiograms [ECGs]), are performed throughout the study. The study hypothesis is that topiramate will improve insulin sensitivity in type 2 diabetic patients and will be well tolerated. Patients will be randomized to receive 192 mg/day (96mg twice daily) of topiramate, or placebo, per mouth for 9 months, with an option of topiramate treatment increasing to 256mg/day both groups during the extension period of 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a history of Type 2 diabetes for 6 months, treated either by diet alone or by sulfonylurea for at least 6 months
* Hemoglobin A1c between 6.5% and 10%
* BMI between 27 and 50
* Non-smokers
* Female patients must be postmenopausal for at least 1 year, surgically incapable of childbearing, practicing an acceptable method of contraception

Exclusion Criteria:

* Unstable endocrine disease
* Significantly abnormal liver function or kidney functions
* History of schizophrenia, major depressive disorder or eating disorder
* History of epilepsy, kidney stones or substance (alcohol) abuse

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2000-04; Study Completion 2002-05 (Actual)

PRIMARY OUTCOMES:
Mean change in insulin sensitivity from baseline to Month 9.

SECONDARY OUTCOMES:
Mean change, baseline to Month 9, in body weight and composition, Body Mass Index (BMI), lipid profile, fasting glucose; blood pressure; safety evaluations (adverse events) during study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A Study of the Safety and Effectiveness of Topiramate on Insulin Sensitivity in Overweight or Obese Patients with Type 2 Diabetes — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=537&filename=CR003715_CSR.pdf